CLINICAL TRIAL: NCT03305835
Title: Characterization of Monogenic Kidney Stone Diseases
Brief Title: Monogenic Kidney Stone - Genetic Testing
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David J. Sas, Principal Investigator, Mayo Clinic
Other Study IDs: 17-005513; U54DK083908 (NIH)
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Rare Kidney Stone Diseases
Keywords: Primary Hyperoxaluria (PH); Hyperoxaluria; PH; PH 1; PH 2; PH 3; Dent Disease; Dent 1; Dent 2; Cystinuria; APRT Deficiency; 24-Hydroxylase Deficiency; CYP24A1
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria; Dent Disease; Cystinuria; Adenine phosphoribosyltransferase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples retained for potential future use, with consent of subjects only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will attempt to identify the specific gene (coded in the DNA) and changes (mutations) within that gene that are the cause of monogenic kidney stone disease. This study will help researchers determine the characteristics of the stone disease associated with specific genes and mutations. This information may help develop more effective treatments for monogenic kidney stone diseases.

DETAILED DESCRIPTION:
Have a blood test (about 2 teaspoons; ½ to 1 teaspoons for children) or buccal cell collection for DNA or RNA isolation • Complete a kidney stone history questionnaire

In addition to the above testing, family members may be asked to participate in the following:

• Complete a 24 hr. urine collection Your samples will undergo genetic testing. We will share the results with your local doctor. All family members, of a patient whose genetic testing showed no known mutations, will not be tested. These samples will be stored for future research.

ELIGIBILITY:
Inclusion Criteria:

Participants meet at least one of the following criteria:

1. Patients <18yrs with a history of kidney stones, and/or nephrocalcinosis, OR
2. Patients >18yrs with a history of kidney stones, and/or nephrocalcinosis and at least one of the following:

   1. Family history of stones or nephrocalcinosis or unexplained kidney failure
   2. Growth retardation
   3. Metabolic bone disease
   4. Unusual stone composition or pathologic or urinary crystals
   5. Proteinuria
   6. Reduced glomerular filtration rate (GFR)
   7. Hypomagnesemia or hypophosphatemia or hypercalcemia
   8. Increased oxalate
   9. Renal cysts, OR
3. Patients with a high clinical suspicion for a monogenic kidney stone disease or a disorder of calcium metabolism OR
4. Patients previously enrolled in the Rare Kidney Stone Consortium 6406 protocol (identified as legacy samples), "Genetic Characterization and Genotype/Phenotype Correlations in Primary Hyperoxaluria." These patients have already consented for their samples to be used in genetic research and that consent will serve to enroll them in this study, OR
5. Patients previously enrolled in the Rare Kidney Stone Consortium 6403 protocol (identified as legacy samples), "Screening for Dent Disease Mutations in Patients with Proteinuria or Hypercalciuria and Calcium Urolithiasis." These patients have already consented for their samples to be used in genetic research and that consent will serve to enroll them in this study, OR
6. Family member of a patient that meets at least one of the above criteria

Exclusion Criteria:

1. Stone formers who do not meet the inclusion criteria for clinical suspicion of one of the monogenic kidney stone diseases
2. Unwilling or unable to provide consent/assent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with clinical characteristics suggestive of monogenic stone disease.
  * Family members of patients with clinical characteristics suggestive of monogenic stone disease.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
symptomatic onset of monogenic stone disease | 5 years
  To identify and define the etiology of monogenic diseases causing nephrolithiasis and nephrocalcinosis by the 90 gene mutation possibly for identification.

SECONDARY OUTCOMES:
Genotype markers | 5 years
  Provide definitive genetic information for research diagnostics by the 90 gene mutation possibly for identification.

CONTACTS AND LOCATIONS:
Overall Officials: David Sas, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Using a limited data set, plans to share data in accordance with NIH funding expectations.

REFERENCES:
- See also: Rare Kidney Stone Consortium — http://www.rarekidneystones.org